CLINICAL TRIAL: NCT03270709
Title: Effect of High-Dose Vitamin D3 on Alveolar Macrophage Function, LL-37, and Oxidative Stress in Smokers and Non-Smokers With and Without HIV
Brief Title: Effect of High-Dose Vitamin D3 in Smokers and Non-Smokers With and Without HIV
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated early due to lack of funding and the COVID-19 pandemic.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jenny Elizabeth Han, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00094833
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: HIV/AIDS; Vitamin D Deficiency; Smoker Lung
Keywords: Vitamin D3; Pulmonary disease; Immunosuppression; HIV; Smoking
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Vitamin D Deficiency; Lung Diseases; Smoking | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: A total of 44 subjects (11 per group, smokers and non-smokers, HIV+, HIV-) will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- HIV+ smokers (Experimental): Vitamin D3 450,000 IU orally
  Interventions: Drug: Vitamin D3 450,000 IU orally
- HIV- non-smokers (Active Comparator): Vitamin D3 450,000 IU orally
  Interventions: Drug: Vitamin D3 450,000 IU orally
- HIV+ non-smokers (Active Comparator): Vitamin D3 450,000 IU orally
  Interventions: Drug: Vitamin D3 450,000 IU orally
- HIV- smokers (Active Comparator): Vitamin D3 450,000 IU orally
  Interventions: Drug: Vitamin D3 450,000 IU orally

INTERVENTIONS:
Drug: Vitamin D3 450,000 IU orally — Study subjects will receive 2 tablets of vitamin D3 for a total of 450,000 IU by mouth.

SUMMARY:
Supplementation with vitamin D improves HIV+ macrophages phagocytosis in vitro. There is evidence to suggest that administering vitamin D can in fact improve immune function in individuals. The study will evaluate the impact of high dose vitamin D in HIV+ smokers' and HIV- smokers' in vivo. The primary goal is to improve innate immune host response to infection in patients already at high risk by virtue of HIV and smoking status.

DETAILED DESCRIPTION:
Tobacco smoke suppresses the lung's ability to fight infection. Smoking is three times more prevalent in the HIV+ compared to HIV- patients. Viral load was found to be significantly increased in HIV+ smokers compared to HIV+ non-smokers, suggesting that smoking enhances HIV-1 viral replication in macrophages, which contributes to disease progression. Vitamin D deficiency has been associated with increased mortality in HIV+ persons, but there is limited research on how this is impacting the health of these highest risk patients and if aggressive repletion with vitamin D can improve overall health.The study team hypothesizes that vitamin D administration will increase pathogen clearance and improve innate immune function.

The proposed pre and post interventional study is designed to characterize alveolar macrophage function and lung immunity according to tobacco use and HIV status, and determine the impact of high dose oral vitamin D3 on AM phagocytic function and innate immunity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects living with HIV-1 infection who have been on anti-retroviral therapy (ART) for a minimum of 12 months and are followed longitudinally for their HIV healthcare;
* Ability to give informed consent.

Exclusion Criteria:

* Age <18 yrs old;
* Known or possible pregnancy or breastfeeding;
* Documented history of cirrhosis or a direct bilirubin ≥ 2.0 mg/dL;
* Documentation of left ventricular ejection fraction < 40% or myocardial infarction within the past 6 months;
* End-stage renal disease requiring dialysis or a serum creatinine ≥ 2 mg/d;
* Spirometry with forced vital capacity (FVC) or forced expiratory volume (FEV1)< 70% of predicted value;
* Bleeding disorders such as thrombocytopenia or significant gastrointestinal bleeding within the past year;
* Inability to undergo bronchoscopy safely;
* High risk behaviors without known HIV status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Difference in alveolar macrophage (AM) phagocytic index between HIV+ smokers compared to HIV- non-smokers. | Day 1 of the study prior to vitamin D administration.
  A phagocytic index will be determined by challenging AM isolated from bronchoalveolar lavage (BAL) to Staph. Aureus in vitro.
Difference in phagocytosis percent positive between HIV+ smokers compared to HIV- non-smokers, prior to vitamin D administration. | Day 1 of the study prior to vitamin D administration.
  Difference in phagocytosis percent positive between HIV+ smokers compared to HIV- non-smokers will be calculated.
Difference in alveolar macrophage (AM) phagocytic index before and after vitamin D administration. | Day 1 of the study prior to vitamin D administration, Day 7 after vitamin D administration
  A phagocytic index will be determined by challenging AM isolated from bronchoalveolar lavage (BAL) to Staph. Aureus in vitro.

SECONDARY OUTCOMES:
Difference in total and free vitamin D (25(OH) D) between HIV+ smokers compared to HIV- non-smokers, prior to vitamin D administration. | Day 1 of the study prior to vitamin D administration.
  Difference in total and free 25(OH) D between HIV+ smokers compared to HIV- non-smokers will be measure by ELISA (enzyme-linked immunosorbent assay) levels.
Difference in peptide LL-37 between HIV+ smokers compared to HIV- non-smokers, prior to vitamin D administration. | Day 1 of the study prior to vitamin D administration.
  Difference in an antimicrobial and immunostimulating/-modulating peptide LL-37 between HIV+ smokers compared to HIV- non-smokers will be calculated.
Difference in tumor necrosis factor alpha (TNF-α) between HIV+ smokers compared to HIV- non-smokers, prior to vitamin D administration. | Day 1 of the study prior to vitamin D administration.
  Difference in tumor necrosis factor alpha (TNF-α) - cytokine involved in systemic inflammation - between HIV+ smokers compared to HIV- non-smokers will be calculated .
Difference in messenger ribonucleic acid (mRNA) expression of LL-37 between HIV+ smokers compared to HIV- non-smokers, prior to vitamin D administration. | Day 1 of the study prior to vitamin D administration.
  Difference in mRNA expression of antimicrobial peptide LL-37 between HIV+ smokers compared to HIV- non-smokers will be calculated.
Difference in alveolar oxidative stress between HIV+ smokers compared to HIV- non-smokers, prior to vitamin D administration. | Day 1 of the study prior to vitamin D administration.
  Difference in alveolar oxidative stress between HIV+ smokers compared to HIV- non-smokers will be measured using AM isolated from bronchoalveolar lavage (BAL) .
Difference in total and free vitamin D (25(OH) D) before and after vitamin D administration. | Day 1 of the study prior to vitamin D administration, Day 7 after vitamin D administration
  Difference in total and free vitamin D (25(OH) D) will be measure by ELISA (enzyme-linked immunosorbent assay)
Difference in peptide LL-37 before and after vitamin D administration. | Day 1 of the study prior to vitamin D administration, Day 7 after vitamin D administration
  Difference in peptide LL-37 levels will be calculated.
Difference in tumor necrosis factor alpha (TNF-α) before and after vitamin D administration. | Day 1 of the study prior to vitamin D administration, Day 7 after vitamin D administration
  Difference in tumor necrosis factor alpha (TNF-α) will be calculated.
Difference in mRNA expression of LL-37 before and after vitamin D administration. | Day 1 of the study prior to vitamin D administration, Day 7 after vitamin D administration
  Difference in mRNA expression of LL-37 will be calculated.
Difference in alveolar oxidative stress before and after vitamin D administration. | Day 1 of the study prior to vitamin D administration, Day 7 after vitamin D administration
  Difference in alveolar oxidative stress will be measured using AM isolated from bronchoalveolar lavage (BAL) .

CONTACTS AND LOCATIONS:
Overall Officials: Jenny E Han, MD, MSc, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Atlanta VA Medical center, Atlanta, Georgia
  - Grady Health System (non-CRN), Grady Health System (CRN), Ponce Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Undecided